CLINICAL TRIAL: NCT05952687
Title: iSTAR: Phase 1b Trial of Idasanutlin and Selinexor Therapy For Children With Progressive/Relapsed Atypical Teratoid Rhabdoid Tumors, Extra-CNS Malignant Rhabdoid Tumors Or Synchronous/Metachronous Rhabdoid Tumors
Brief Title: Trial of Idasanutlin and Selinexor Therapy for Children With Progressive/Relapsed AT/RT or Extra-CNS Malignant Rhabdoid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug withdrawn by company.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iSTAR; NCI-2023-05552 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Rhabdoid Tumor; Atypical Teratoid/Rhabdoid Tumor; Atypical Teratoid/Rhabdoid Tumor of CNS; CNS Tumor
MeSH Terms: conditions — Rhabdoid Tumor; Central Nervous System Neoplasms | interventions — RG7388; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Finding/Safety Phase (Experimental): Patients with progressive/relapsed atypical teratoid/rhabdoid tumors (AT/RT) & malignant rhabdoid tumors (MRT) or synchronous/metachronous AT/RT &MRT
  Interventions: Drug: Idasanutlin; Drug: Selinexor
- Expansion Phase: Stratum A (Experimental): Patients with progressive/relapsed AT/RT
  Interventions: Drug: Idasanutlin; Drug: Selinexor
- Expansion Phase: Stratum B (Experimental): Patients with progressive/relapsed MRT
  Interventions: Drug: Idasanutlin; Drug: Selinexor
- Expansion Phase: Stratum C (Experimental): Patients with progressive/relapsed, synchronous/metachronous AT/RT & MRT
  Interventions: Drug: Idasanutlin; Drug: Selinexor

INTERVENTIONS:
Drug: Idasanutlin — Patients will receive idasanutlin dosed once daily on Days 1-5 of a 28-day cycle starting with 80% of the RP2D determined in the ongoing pediatric iMATRIX trial using single agent idasanutlin.
  Other Names: RO5503781
  Arms: Dose Finding/Safety Phase
Drug: Idasanutlin — Patients will receive idasanutlin dosed once daily on Days 1-5 of a 28-day cycle starting with the RP2D determined in the dose-finding/safety phase.
  Other Names: RO5503781
  Arms: Expansion Phase: Stratum A; Expansion Phase: Stratum B; Expansion Phase: Stratum C
Drug: Selinexor — Patients will receive selinexor on Day 4 of each of the first 3 weeks of a 28-day cycle. Selinexor will be skipped on week 4 of each cycle.
  Other Names: KPT-330

SUMMARY:
iSTAR is an open-label, multi-center, phase 1b study of oral XPO1 inhibitor selinexor and oral MDM2 inhibitor idasanutlin in children with progressive or recurrent atypical teratoid/rhabdoid tumors (AT/RT), malignant rhabdoid tumors (MRT) and synchronous/metachronous rhabdoid tumors.

Primary Objectives

* To determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of combination treatment with oral idasanutlin and selinexor in children with recurrent or progressive AT/RT or MRT.
* To characterize the plasma pharmacokinetics of oral idasanutlin and selinexor in children with recurrent or progressive AT/RT or MRT, to assess potential covariates to explain the inter- and intra-individual pharmacokinetic variability.

Secondary Objectives

* Evaluate safety of the combination treatment with oral idasanutlin and selinexor in children
* Evaluate efficacy of the combination treatment of idasanutlin and selinexor as measured by objective response (partial response [PR] or complete response [CR]) rate separately in progressive/relapsed AT/RT and progressive/relapsed MRT
* Estimate progression-free and overall-survival separately in progressive/relapsed AT/RT and progressive/relapsed MRT

DETAILED DESCRIPTION:
Patients will receive idasanutlin dosed once daily on Days 1-5 of a 28-day cycle starting with 80% of the RP2D determined in the ongoing pediatric iMATRIX trial (NCT04029688) using single agent idasanutlin. Patients will receive selinexor on Day 4 of each of the first 3 weeks of a 28-day cycle. Selinexor will be skipped on week 4 of each cycle.

The dose-finding/safety phase will test two dosing frequencies and two dose levels of selinexor [100, and 75% of the RP2D from the COG trial (NCT02323880)] using single agent selinexor and 2 dose levels of idasanutlin [80% and 100% of the RP2D from the pediatric single agent idasanutlin iMATRIX study (NCT04029688)]. In the COG trial, ADVL1414, the RP2D of single agent selinexor was 35mg/m2 administered weekly of a 28-day cycle without any break. In our trial we propose to skip selinexor during week 4 (dose levels 1). If unexpected toxicity is encountered in dose level 1, St. Jude will open dose level -1(reduced frequency of selinexor dosing) and dose level -2 (reduced dose and frequency of selinexor dosing). However, if dose level 1 is well tolerated, then the St. Jude will open dose level 2 for enrollment (100% of RP2D of single agent selinexor and idasanutlin).

Once the RP2D is established, patients enrolled on the dose-finding/safety phase at this dose level will continue treatment and will be included in the response analysis in the expansion stage. Those patients who are enrolled on the dose-finding/safety phase at a lower dose level and are still on treatment will have their doses optimized following determination of the RP2D. Patients may continue treatment for a maximum of 2 years, or 26 cycles, in absence of progressive disease.

ELIGIBILITY:
Inclusion Criteria: Screening Phase, All Participants

* Participant and/or guardian can understand and will sign a written informed consent document according to institutional guidelines.
* Before patient screening and registration, written informed consent, also concerning data and sample transfer, must be given according to ICH/GCP and national/local regulations
* Children, adolescents, and young adults with relapsed/progressive AT/RT, MRT, or synchronous/metachronous rhabdoid tumor that is histologically confirmed by the enrolling institution. Patients must have failed at least one frontline therapy other than surgery to be eligible.
* Age at enrollment ≥ 6 months to 25 years
* Tumor sample is available from the time of diagnosis or relapse. If tumor sample is not available for deposition but molecular analysis was performed using a non-INFORM registry or non-CLINGEN molecular pipeline, transfer of molecular data (DNA methylation, whole exome and RNA sequencing) must be completed prior to enrollment. However, these tests will have to be completed in a CLIA certified facility.
* Patient has fully recovered from the acute toxic effects of chemotherapy, immunotherapy, or radiation therapy or is anticipated to do so prior to enrolling on this study:

  * Myelosuppressive chemotherapy: patient has not received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (4 and 6 weeks if prior temozolomide and nitrosourea, respectively).
  * Hematopoietic growth factors: at least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim or biosimilar growth factor.
  * Biologic anti-neoplastic agent (except monoclonal antibodies): at least 7 days must have elapsed since completion of therapy with a biologic agent prior to enrollment. For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the 7 days, during which adverse events are known to occur, up to a maximum of 30 days prior to initiation of study treatment.
  * Monoclonal antibodies: Thirty days or at least three half-lives must have elapsed since prior therapy that included a monoclonal antibody, whichever is later prior to initiation of study treatment.
  * Treatment with cellular therapy (e.g., CAR-T cell infusion) for anti-neoplastic intent within 30 days prior to initiation of study treatment
  * Radiation therapy: at least 3 months must have elapsed since any previous irradiation to the site of disease prior to study enrollment, unless measurable disease is confirmed by biopsy or is present at a site separate from the irradiated area or meets CSF criteria for enrollment

Inclusion Criteria: Dose-Finding/Safety Phase and Expansion Phase

* Disease that is measurable as defined by RAPNO criteria or RECIST v1.1 (as appropriate). A patient who has no measurable disease will be allowed to enroll if one of the following criteria is met:

  * there is evidence of leptomeningeal disease
  * CSF presence of tumor cells by cytology confirmed on 2 separate occasions at least 1 week apart.
* Adequate performance status:

  * Patients <16 years of age: Lansky ≥50%
  * Patients ≥16 years of age: Karnofsky ≥50%
  * Transient states like infections can be accepted, stable disabilities resulting from disease/surgery (posterior fossa syndrome, hemiparesis, amputations, etc.) can be accepted and will not be considered for Lansky/ Karnofsky assessments.
* Stable neurologic deficits on a stable dose of corticosteroids (if applicable) for at least 1 week before study enrollment.
* Patient can swallow oral study medication or should have a nasogastric for minimum size of the NG tube that may be used) or G-tube for the administration of the medication.
* Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment.
* For females of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse or use contraception, agreement to refrain from donating eggs
* For males: agreement to remain abstinent (refrain from heterosexual intercourse or use a condom, and agreement to refrain from donating sperm
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* No prior therapy with the combination of MDM2 inhibitors and XPO1 inhibitors.
* Adequate end-organ function defined by the following laboratory results obtained within 14 days prior to initiation of study drug:

  * Bone marrow function: normal bone marrow function as defined by:

    * a hemoglobin concentration >8 g/dL (with or without support);
    * absolute neutrophil count (ANC) > 1,000/mm3, and
    * platelet count >75,000/ mm3 (unsupported for 72 hours)
  * Adequate renal function as defined by CrCl ≥60 mL/min/1.73 m2
  * Adequate liver function as defined by alanine aminotransferase (ALT) and aspartate aminotransferase (AST) concentration ≤ 3 x upper limit of normal (ULN) per institutional practice and total bilirubin ≤ 1.5 × ULN for age. Serum albumin ≥ 2 g/dL
  * Adequate Pancreatic Function defined as:

    * Serum amylase ≤ 1.5 x ULN as per institutional practice
    * Serum lipase ≤ 1.5 x ULN as per institutional practice
* Adequate cardiac function as defined by:

  * ECG with normal QTc interval < 450 ms as determined by Fridericia correction
  * Fractional shortening (FS) ≥28% or left ventricular ejection fraction (LVEF) ≥50% as determined by echocardiography or multigated acquisition scan (MUGA)within 28 days prior to initiation of study therapy.

    * Depending on institutional standard, either FS or LVEF is adequate for enrollment if only one value is measured; if both values are measured, then both values must meet the above criteria.
* Life expectancy ≥ 3 months, in the investigator's judgment

Exclusion Criteria: Screening Phase

* Significant nausea and vomiting (CTCAEv5 grade 3 or more), chronic diarrhea, malabsorption despite maximal supportive care or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies). Known active hepatitis B (e.g., hepatitis B surface antigen reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to study treatment. Patients with a known history of hepatitis C virus infection and positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Clinically significant, uncontrolled heart disease.
* Pregnant or lactating women at the time of enrollment.

Exclusion Criteria Dose Finding/Safety Phase and Expansion Phase, All Cohorts

* Major surgery within 21 days of the first dose or anticipate need for major surgical procedure during the cycle of the study. Gastrostomy tube placement, ventriculo-peritoneal shunt, ommaya reservoir placement, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery
* Myeloablative therapy with autologous hematopoietic stem cell rescue within 30 days or allogeneic hematopoietic stem cell rescue within 100 days of study treatment initiation
* Received the following within 7 days prior to initiation of study treatment

  * Strong CYP2C8 inhibitors
  * CYP2C8 substrates
  * OATP1B1/3 substrates
* Received strong CYP2C8 and strong CYP3A4 inducers within 14 days prior to the initiation of study treatment
* Patients unable to temporarily interrupt treatment with oral or parenteral anticoagulants/anti-platelet agents (e.g., warfarin, chronic daily treatment with aspirin [> 325 mg/day], clopidogrel, dabigatran, apixaban, rivaroxaban) during the treatment phase. These agents must be discontinued 7 days (or 5 half-lives), whichever is longer prior to the start of study medication.
* Infection considered by the investigator to be clinically uncontrolled or of unacceptable risk to the patient upon induction of neutropenia, including patients who are, or should be on antimicrobial agents for the treatment of active infection such as the following:

  * Fungal infection other than mucosal candidiasis, within <2 weeks of completing appropriate systemic antifungal therapy
  * Bacterial infection with positive cultures in the 7 days prior to dosing
  * Patients who have received <5 days of appropriate antibiotic or antiviral therapy for an identified infection
  * Neutropenic fever considered infection-related within 72 hours prior to dosing
  * History of symptomatic Clostridium difficile (C. diff infection that has since resolved and patient has normal stool consistency and frequency and/or a negative C diff stool test.
* Biopsy confirmed radiation therapy induced pseudoprogression in CNS tumors
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Should not be receiving any other anti-cancer treatment.
* Pregnant or breastfeeding females, or intending to become pregnant during the study
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 28 weeks after stopping study therapy are not eligible.
* Presence of any CTCAE ≥ Grade 2 acute clinically significant treatment-related toxicity with the exception of alopecia, ototoxicity, peripheral neuropathy and parameters otherwise permitted in the inclusion criteria (e.g. hematological criteria)

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of combination treatment with oral idasanutlin and selinexor in children with recurrent or progressive AT/RT or MRT in the dose finding/safety phase. | 1 month after start of idasanutlin and selinexor treatment
  The MTD is empirically defined as the highest dose level at which six patients have been treated with at most one patient experiencing a DLT and the next higher dose level has been determined to be too toxic. The MTD estimate will not be available if the lowest dose level studied is too toxic or the highest dose level studied is considered safe. In the latter case, the highest studied safe dose may be considered at the recommended phase 2 dose (RP2D). The MTD estimate will be limited to evaluable patients and toxicity assessments from course 1 (28 days). The RP2D will be based on the MTD and the totality of the safety/efficacy data.
Idasanutlin plasma apparent systemic clearance (CL/F) in children with recurrent or progressive AT/RT or MRT | 1 month after start of idasanutlin and selinexor treatment
  For each patient, idasanutlin plasma concentration-time data will be analyzed using non-compartmental methods to estimate the plasma CL/F.
Idasanutlin area under the plasma concentration time curve (AUC) in children with recurrent or progressive AT/RT or MRT | 1 month after start of idasanutlin and selinexor treatment
  For each patient, idasanutlin plasma concentration-time data will be analyzed using non-compartmental methods to estimate the AUC.

SECONDARY OUTCOMES:
Objective response rate in subjects with progressive/relapsed AT/RT | Approximately 2 years from start of treatment
  An objective response is defined as a partial or complete response. Response must be at least a partial response in patients with measurable disease and at least a complete response in patients with evaluable disease and must be sustained for approximately 8 weeks (the time of the next regularly scheduled imaging assessment). The objective response rate will be reported with a 95% confidence interval.
Objective response rate in subjects with progressive/relapsed MRT | Approximately 2 years from start of treatment
  An objective response is defined as a partial or complete response. Response must be at least a partial response in patients with measurable disease and at least a complete response in patients with evaluable disease and must be sustained for approximately 8 weeks (the time of the next regularly scheduled imaging assessment). The objective response rate will be reported with a 95% confidence interval.
Progression-free survival in subjects with progressive/relapsed AT/RT | Approximately 7 years from start of treatment
  Progression-free survival is defined as the interval of time between date of initiation of protocol treatment and date of documentation of progression of disease (PD), death due to any cause, or date of last follow-up. Progression-free survival will be estimated using the method of Kaplan and Meier.
Progression-free survival in subjects with progressive/ relapsed MRT | Approximately 7 years from start of treatment
  Progression-free survival is defined as the interval of time between date of initiation of protocol treatment and date of documentation of progression of disease (PD), death due to any cause, or date of last follow-up. Progression-free survival will be estimated using the method of Kaplan and Meier.
Overall survival in subjects with progressive/relapsed AT/RT | Approximately 7 years from start of treatment
  OS is defined as the interval of time between date of diagnosis and date of death due to any cause or date of last follow-up. Overall survival will be estimated using the method of Kaplan and Meier.
Overall survival in subjects with progressive/ relapsed MRT | Approximately 7 years from start of treatment
  OS is defined as the interval of time between date of diagnosis and date of death due to any cause or date of last follow-up. Overall survival will be estimated using the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Principal Investigator — St. Jude Children's Research Hospital

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042...